CLINICAL TRIAL: NCT01601197
Title: A Study of Two Injection Techniques Added to Proven Strategies to Reduce Pain in One- to Twelve-month Old Infants Undergoing Immunization
Brief Title: A Study of Two Injection Techniques to Reduce Pain in Infants Undergoing Immunization
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Associate Professor, Leslie Dan Faculty of Pharmacy, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27518
Record Dates: First submitted 2012-05-13; First posted 2012-05-17 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Infants; Immunization; Pain Management
Keywords: immunization; pain management; infants; tactile stimulation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tactile stimulation (Experimental): Ipsilateral limb will be rubbed immediately before, during and after immunization injection(s)
  Interventions: Behavioral: Tactile stimulation
- No tactile stimulation (No Intervention): There will be no tactile stimulation of ipsilateral limb before, during and after immunization injection(s)

INTERVENTIONS:
Behavioral: Tactile stimulation — Immunizer will rub the ipsilateral limb before, during and after immunization injection(s)
  Arms: Tactile stimulation

SUMMARY:
Immunization injections are a significant source of pain for infants. Tactile stimulation (rubbing/applying pressure) may be an effective and feasible pain-relieving intervention - it is cost neutral, and has been shown to be effective in children and adults undergoing injections. The aim of this study is to determine the added benefit of tactile stimulation when added to other proven analgesic interventions during routine infant immunization injections.

DETAILED DESCRIPTION:
Immunization injections are a significant source of pain for infants. At present, effective and feasible pain-relieving interventions include sugar water, fast injection without aspiration, and holding infants during the procedure. These methods, however, do not eliminate pain in all infants. Additional interventions are therefore needed.

Tactile stimulation (rubbing/applying pressure) has been shown to reduce injection pain in children and adults, and may be a suitable intervention for infant injections. It is cost neutral, requires no preparation, and is easily incorporated into practice.

The aim of this study is to determine the effectiveness of tactile stimulation when added to other proven analgesic interventions on reducing pain during infant immunization injections.

ELIGIBILITY:
Inclusion Criteria:

* infants 1-12 months of age receiving routine immunization injections in an outpatient pediatric clinic in Toronto

Exclusion Criteria:

* impaired neurological development
* history of seizure
* use of topical anesthetics
* use of sedatives or narcotics within 24 hours
* fever or illness that would prevent administration of vaccine
* prior participation in the trial

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Infant Pain as assessed by the Modified Behavioral Pain Scale | First 15 seconds after injection
  assessed from videotaped procedure

SECONDARY OUTCOMES:
Parent rating of infant pain using the Numerical Rating Scale | first minute after injection
Immunizer rating of infant pain using the Numerical Rating Scale | first minute after injection
Infant crying time | duration of crying after injection
  assessed from videotaped procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — Leslie Dan Faculty of Pharmacy, University of Toronto, 144 College Street, Toronto, Ontario M5S 3M2 Canada
Locations (1):
- Dr. Tommy Ho Pediatric Clinic, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Taddio A, Ho T, Vyas C, Thivakaran S, Jamal A, Ilersich AF, Hogan ME, Shah V. A randomized controlled trial of clinician-led tactile stimulation to reduce pain during vaccination in infants. Clin Pediatr (Phila). 2014 Jun;53(7):639-44. doi: 10.1177/0009922814526976. Epub 2014 Mar 14. PMID 24634424